CLINICAL TRIAL: NCT05838508
Title: Effect of Physical Activity Pattern on Cardiometabolic Health
Acronym: PACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jingyi Qian, Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023P001025; R00HL148500 (NIH)
Record Dates: First submitted 2023-04-07; First posted 2023-05-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Life Style
Keywords: exercise; circadian system; physical activity; glucose tolerance; blood pressure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise A-B Intervention (Experimental): The Exercise A first, then the Exercise B intervention.
  Interventions: Behavioral: Exercise intervention
- Exercise B-A Intervention (Experimental): The Exercise B first, then the Exercise A intervention.
  Interventions: Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Exercise intervention — Research participants will be assigned to two exercise conditions.

SUMMARY:
The goal of this study is to understand the interaction between the circadian system and physical activity.

Participants will:

* complete 2 inpatient stays
* perform moderate exercise
* be provided with identical meals
* have frequent blood draws
* provide urine and saliva samples

DETAILED DESCRIPTION:
The endogenous circadian system (i.e., an internal biological rhythm) plays an important role in regulating blood glucose, blood pressure, and energy expenditure. Physical activity improves health and reduces the risk for cardiovascular diseases and type 2 diabetes. The goal of this study is to understand the interaction between the circadian system and physical activity. We aim to test whether such relationship between the circadian system and physical activity can be used to enhance the health benefits of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 yr old
* Body mass index (BMI) 18.5 - 34.9 kg/m2
* No acute, chronic or debilitating medical conditions (e.g. metabolic, cardiovascular, respiratory, neurological, cancers, etc.)
* Willing to adhere to the protocol requirements for the duration of the study

Exclusion Criteria:

* Currently smoking/vaping or 5 or more years of smoking/vaping
* Currently pregnant or breastfeeding
* History of drug or alcohol dependency
* History of psychiatric illness or disorder
* Any hospitalization due to COVID-19
* Inability to exercise for any reason
* Any known contraindication to exercise testing based on current ACSM guidelines

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
glucose level | 24-hour test period after exercise
  mean glucose level after exercise session
mean arterial pressure | 24-hour test period after exercise
  mean arterial pressure after exercise session

SECONDARY OUTCOMES:
insulin sensitivity index | about 12 and 24 hours after exercise
  Oral Minimal Model method estimates mean insulin sensitivity based on blood glucose and insulin levels from two mixed meal tests after exercise session
beta-cell function index | about 12 and 24 hours after exercise
  Oral Minimal Model method estimates mean beta-cell function based on blood glucose, insulin and c-peptide levels from two mixed meal tests after exercise session
total peripheral resistance | 24-hour test period after exercise
  total peripheral resistance derived from BP waveform measured by finger plethysmography
autonomic nervous system activity | 24-hour test period after exercise
  derived by time-domain heart rate variability analysis

OTHER OUTCOMES:
resting energy expenditure | 24-hour test period after exercise
  energy expenditure will be measured at 1-2 hours interval by indirect calorimetry
respiratory exchange ratio | 24-hour test period after exercise
  respiratory exchange ratio will be measured at 1-2 hours interval by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Qian, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No